CLINICAL TRIAL: NCT06275152
Title: The Protective Effect of Remote Ischemic Conditioning on Residual Renal Function in Hemodialysis Patients: A Multicenter, Randomized, Double-blind, Sham-controlled Trial.
Brief Title: The Protective Effect of Remote Ischemic Conditioning on Residual Renal Function in Hemodialysis Patients (RIC-HD)
Acronym: RIC-HD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Yuanjun Yang (Other)
Responsible Party: Sponsor-Investigator, Yuanjun Yang, Director, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HDRIC-01
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: End-stage Renal Disease
Keywords: Hemodialysis; residual renal function; Remote ischemic conditioning
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Intervention Model Description: randomized controlled pilot study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Only Research Assistant will be unblinded. Participant, clinical team, PI, etc. will all be blinded to the randomization group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIC group (Experimental): RIC interventions will be applied to the upper extremity for a total of 20 cumulative minutes of limb ischemia, at a pressure of 200 mmHg.
  Interventions: Device: Remote ischemic conditioning
- Sham Remote Ischemic Conditioning (Sham Comparator): The sham-RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Interventions: Device: Sham Remote Ischemic Conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — RIC is a non-invasive therapy that performed by an electric auto-control device with cuff placed on arm. RIC procedure during which bilateral arm cuffs are inflated to a pressure of 200mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: RIC group
Device: Sham Remote Ischemic Conditioning — The sham-RIC procedure during which bilateral arm cuffs are inflated to a pressure of 60mmHg for five cycles of 5 min followed by 5 min of relaxation of the cuffs.
  Arms: Sham Remote Ischemic Conditioning

SUMMARY:
Hemodialysis (HD) is the main renal replacement therapy for patients with end-stage renal disease. However, factors such as hemodynamic instability can lead to gradual loss of residual renal function (RRF) in HD patients. The loss of RRF not only affects the adequacy of dialysis and complications control but also impacts the patients' quality of life and survival. Unfortunately, there are currently no effective methods to protect RRF. The purpose of this study is to validate the protective effect of remote ischemic conditioning (RIC) on RRF in HD patients. This will provide evidence for the application of RIC in protecting RRF in HD patients.

DETAILED DESCRIPTION:
Hemodialysis (HD) is the main renal replacement therapy for patients with end-stage renal disease. However, factors such as hemodynamic instability can lead to gradual loss of residual renal function (RRF) in HD patients. The loss of RRF not only affects the adequacy of dialysis and complications control but also impacts the patients' quality of life and survival. Unfortunately, there are currently no effective methods to protect RRF. Remote ischemic conditioning (RIC) is a simple, safe, non-invasive, and non-pharmacological intervention. It induces the remote organs to develop an anti-ischemic injury capacity through repeated and brief ischemic stimuli on limbs, thereby reducing ischemic damage. RIC is a clinically feasible method that is easy to implement and promote. It has been widely used in the treatment and research of cardiovascular and cerebrovascular diseases, as well as in the prevention of acute kidney injury related to thoracoabdominal surgery and contrast agents. Studies have also found that RIC significantly reduces myocardial ischemic injury in HD patients. Theoretically, RIC can also be used to protect the RRF in HD patients. This study aims to validate the protective effect of RIC on RRF in HD patients. This will provide evidence for the application of RIC in protecting RRF in HD patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* First-time initiators of hemodialysis treatment for end-stage renal disease patients;
* Urine output > 500ml/day or GFR > 3ml/min/1.72m2;
* Hemodialysis access as a central venous catheter.
* Signed and dated informed consented is obtained;

Exclusion Criteria:

* Active infection;
* Infectious disease;
* Expected dialysis duration < 6 months;
* Presence of vascular access dysfunction (blood flow rate < 180ml/min);
* Patients who had contraindication of remote ischemic conditioning, such as severe soft tissue injury, fracture or vascular injury in the upper extremities, venous thrombosis in the acute or subacute stage of upper extremities;
* Pregnancy or lactation women;
* Patients who are participating in other clinical studies, or who have participated in other clinical studies within 3 months prior to enrollment;
* Unwillingness to be followed up or poor adherence to treatment;
* Other circumstances that the investigator considers unsuitable for enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02-20 (Estimated); Primary Completion 2026-01-19 (Estimated); Study Completion 2026-01-19 (Estimated)

PRIMARY OUTCOMES:
time to anuria | 10 months
  defined as ≤100 ml/d or ≤200 ml of urine volume in the short interdialytic period
residual renal function (RRF) | 10 months
  The RRF was calculated from an interdialytic urine collection and pre- and post-dialysate blood samples as the mean of the urea and creatinine clearances adjusted for body surface area using a "GFR calculator"
Change in the renal cerebral oxygen saturation | 10 months
  Measured by Near Infrared Spectroscopy

SECONDARY OUTCOMES:
serum creatinine | 10 months
  Taking a blood test to evaluation creatinine
serum urea nitrogen | 10 months
  Taking a blood test to evaluation urea nitrogen
C-reactive protein (CRP) | 10 months
  Taking a blood test to evaluation CRP
Interleukin-6 | 10 months
  Taking a blood test to evaluation Interleukin-6
TFF3 | 10 months
  Taking a urine test to evaluation TFF3
KIM-1 | 10 months
  Taking a urine test to evaluation KIM-1
IP-10 | 10 months
  Taking a urine test to evaluation IP-10

OTHER OUTCOMES:
hemoglobin | 10 months
  Collect data at baseline and during each follow-up visit.
systolic pressure | 10 months
  Collect data at baseline and during each follow-up visit
diastolic pressure | 10 months
  Collect data at baseline and during each follow-up visit.

CONTACTS AND LOCATIONS:
Overall Officials: Guangyan Cai, Study Director — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China